CLINICAL TRIAL: NCT02523768
Title: Prevention in Recipients With Primary IgA Nephropathy of Recurrence After Kidney Transplantation: ATG-F Versus Basiliximab as Induction Immunosuppressive Treatment
Acronym: PIRAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties for recruting patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0908143; 2009-018189-36 (EudraCT Number); A100405-32 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-04; First posted 2015-08-14 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Glomerulonephritis; IgAN
MeSH Terms: conditions — Glomerulonephritis | interventions — Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG-F (Experimental): The ATG-Fresenius® is administered by slow infusion over four hours after antihistamine (2 bulbs Polaramine® IV) and intravenous methylprednisolone (minimum 30mg); it is started on day 0 prior to surgery at doses of 4 mg / kg, and then continued to day 1, day 2 to 4mg / kg, then day 3, day 4 at the dose of 3 mg / kg
  Interventions: Drug: ATG-F
- Simulect (Active Comparator): The anti CD25 (basiliximab, Simulect®) is administered intravenously before surgery of renal transplantation (Day 0 and Day + 4 (1 ampoule of 20 mg x 2 times).
  Interventions: Drug: Simulect

INTERVENTIONS:
Drug: ATG-F
  Arms: ATG-F
Drug: Simulect
  Arms: Simulect

SUMMARY:
IgA nephropathy (IgAN) is a histologically defined glomerulonephritis (renal biopsy) by the presence of deposits immunoglobulin A (IgA) in the renal mesangium (at least 1+) by immunofluorescence. The clinic allows excluding secondary forms (10-15%). Recurrence of this condition on the renal graft is time-dependent and confirmed in 25 to 50% of 10 years post-transplant.

The primary immunosuppressive induction regimens currently used in kidney transplantation are the anti-lymphocyte globulin (GAL) whose main target is human T lymphocytes (ATG, polyclonal) and monoclonal anti-CD25 antibodies (α chain of the interleukin receptor 2 in the surface of T lymphocytes). Due to their potent and prolonged immunosuppressive properties, the ATG may prevent or delay the recurrence on renal transplant.

The aim of this study was to evaluate the influence of induction therapy (ATG versus Basiliximab) in the cumulative incidence at 5 years of (IgAN) recurrence after a first kidney transplant.

This is a prospective, multicenter, randomized, open trial with a follow-up period of 5 years old.

Patients in the ATG arm will receive 5 antilymphocyte globulin infusions Fresenius® (rabbit immunoglobulin antilymphocyte human T-Fresenius® said ATG) from Day 0 to Day + 4 post-transplant (day 0 one dose of 4mg / kg, day 1 one dose of 4mg/kg, day2 one dose of 4mgkg, day 3 one dose of 3 m/kg and day 4 and one final dose of 3 mg/kg) and the patients in the anti-CD25 arm will receive 2 doses of 20 mg of basiliximab (Simulect®) pn day 0 and day 4 after the graft. The maintenance immunosuppressive therapy is left to the discretion of the center.

The primary endpoint will be the clinical and histological recurrence of IgAN defined by the presence of mesangial deposits of IgA (at least 1) by immunofluorescence on a biopsy of the graft triggered by the onset of proteinuria 1g/j and/or microalbuminuria greater than 300 mg / day.

ELIGIBILITY:
Inclusion Criteria:

* Free, informed, express and written.
* Diagnosis of native kidney primary IgA glomerulonephritis biopsy-proven
* First kidney transplantation (one kidney)

Exclusion Criteria:

* Panel Reactive Antibody (PRA PRA global or class I or class II PRA) over 50% on a serum before transplantation
* Multi-organ graft
* Transplants using donor limits or sub-optimal: donor age ≥ 70 years, donors in the study BIGRAS or taken heart beating donors (tested on computer infusion) or other restriction factors
* IgA glomerulonephritis secondary to HSP (Henoch-Schonlein purpura) or Systemic Lupus Erythematosus (SLE) or alcoholic cirrhosis
* History of cancer older than 5 years or with advanced cancer, but except for non-recurrent skin cancers
* Infectious diseases scalable: tuberculosis, HIV, Hepatitis B virus or Hepatitis C virus infection with viral replication and / or chronic hepatitis
* Allergy to rabbit proteins
* Severe thrombocytopenia (<50,000 platelets/ul)
* Bacterial infection, viral and fungal uncontrolled therapeutically
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-01-08 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
clinical recurrence | 5 years
  onset of proteinuria 1g / j and / or microalbuminuria greater than 300 mg / day
histological recurrence | 5 years
  histological recurrence defined by the presence of mesangial deposits of IgA (at least 1+) by immunofluorescence on a biopsy of the graft

CONTACTS AND LOCATIONS:
Overall Officials: Francois BERTHOUX, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (15):
- France (15):
  - CHU de BESANCON, Besançon
  - CHU de BORDEAUX, Bordeaux
  - Chu Kremlin Bicetre, Le Kremlin-Bicêtre
  - Hopital Edouard HERRIOT, Lyon
  - CHU de MONTPELLIER, Montpellier
  - CHU de NANCY, Nancy
  - CHU de NANTES, Nantes
  - CHU de NICE, Nice
  - Hopital Pitie Salpetriere, Paris
  - Hopital Tenon, Paris
  - Hopital LYON Sud, Pierre-Bénite
  - CHU de SAINT-ETIENNE, Saint-Etienne
  - CHU de STRASBOURG, Strasbourg
  - CHU de TOULOUSE, Toulouse
  - CHRU de TOURS, Tours

IPD SHARING:
Plan to Share IPD: No